CLINICAL TRIAL: NCT05157152
Title: Elevated Liver Enzymes as a Predictor of Acute Kidney Injury in Hospitalized Patients With COVID-19
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Karam Helmy, Resident doctor at internal medicine department, sohag university hospital, Sohag University
Other Study IDs: Soh-Med-21-12-10
Record Dates: First submitted 2021-12-12; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Liver enzymes, serum creatinine, CBC, PCR
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In critically ill patients, AKI is a common complication of COVID-19 infection, occurring in 23% to 43% of cases, and was correlated with poor clinical outcomes.

An increase in liver function tests ( LFTs) has been found in patients with COVID-19 ranging 14%-75% Some studies found higher levels of transaminases in patients with severe COVID-19 pneumonia and in patients dying for COVID-19.

Initial reports indicate a high incidence of abnormal liver tests and acute kidney injury (AKI) in the novel coronavirus infection (COVID-19).

We hypothesis that there is a relationship between COVID-19 patients who are critically ill, liver enzymes and level of serum creatinine

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) affects multiple organ systems and imparts significant morbidity and mortality [1]. Approximately 5% to 14% of patients affected with SARS-CoV-2 will become critically ill [2-4]. While coronavirus disease 2019 (COVID-19) generally begins as a respiratory tract infection, it can damage any organ system. Thus, to improve outcomes, clinicians should search actively for multi-organ involvement to guide appropriate early management [5].

Among affected organs, the kidney is particularly susceptible to COVID-19. Indeed, SARS-CoV-2 has been shown to share the same functional receptor, angiotensin-converting enzyme 2 (ACE2), with a wide variety of organs (such as lung, heart, kidney) [6]. SARS-CoV-2 initiates its infection process by binding to functional receptors on the membrane of a host cell. Postmortem examination of COVID-19 patients revealed varying degrees of acute tubular necrosis, lymphocytic infiltration, and viral RNA, suggesting direct invasion of kidney tubules [7]. In addition to direct kidney damage by the virus, acute kidney injury (AKI) can occur through several proposed mechanisms including acute tubular necrosis induced by sepsis, hypoxia, hypoperfusion, rhabdomyolysis, nephrotoxic drugs, etc.

In critically ill patients, AKI is a common complication of COVID-19 infection, occurring in 23% to 43% of cases, and was correlated with poor clinical outcomes. AKI was defined as per Kidney Disease Improving Global Outcomes (KDIGO) criteria: a change in the serum creatinine of 0.3 mg/dL over 48 h period or 50% increase in baseline creatinine.

An increase in liver function tests ( LFTs) has been found in patients with COVID-19 ranging 14%-75% Some studies found higher levels of transaminases in patients with severe COVID-19 pneumonia and in patients dying for COVID-19.

The clinical relevance of LFTs abnormalities has been controversial, with some studies suggesting its association with the severity of COVID-19 pneumonia, whereas others not.Some limitations affected those studies involving the lack of information about concomitant or previous use of hepatotoxic drugs among the others.

Initial reports indicate a high incidence of abnormal liver tests and acute kidney injury (AKI) in the novel coronavirus infection (COVID-19). However, outcomes in hospitalized patients with COVID-19 and elevated aspartate transaminase (AST) and alanine transaminase (ALT) levels at admission and their associations with AKI are not well understood.

Aim of the work

The aim of this study is to investigate the incidence of liver injury at admission and its contribution to the development of AKI, severity of COVID-19 and outcomes in Sohag University hospital

Patients and methods

Type of the Study:

A prospective, observational cohort study will be conducted between December 2021 and May 2022 among hospitalized COVID-19 patients in Sohag University Hospital.

Patients:

Inclusion criteria :

Patients who are positive for COVID-19 infection in Sohag University Hospital whose ages < 18 years old. (confirmed by polymerase chain reaction (PCR) from nasopharyngeal or oropharyngeal samples) who developed AKI at time of admission or during admission.

Exclusion criteria :

Patients whose ages >18 years old.

Methods A prospective, observational cohort study will be conducted between December 2021 and April 2022 among hospitalized COVID-19 patients in Sohag University Hospital.

The routine laboratory parameters will be measured before the beginning of this Study After conducting a complete physical examination.

demographic, clinical, radiological and laboratory data will be collected at admission. Information on medical history, including comorbidities, symptoms of infection and drugs taken in the previous 14 days before admission will be collected. Vital signs (respiratory rate [RR], body temperature [BT], arterial blood pressure, heart rate [HR], pulse oxygen saturation [SatO2] were collected. Laboratory tests including alanine aminotransferase (ALT), aspartate aminotransferase (AST), serum Albumin, Total protein, serum creatinine, Blood urea nitrogen, serum electrolytes and bilirubin were collected at admission and every 7 ± 2 days during the admission.

Patients diagnosed with COVID-19 will be divided into three groups as mild, moderate, and severe disease to evaluate the relationship between disease severity and AKI. Patients with clinical signs of pneumonia (fever, cough, dyspnoea, fast breathing) plus one of the following: respiratory rate >30 breaths/min; severe respiratory distress;or SpO2 < 90% on room air will be considered as severe cases.

Patients with pneumonia and have no above severity criteria will be considered as moderate cases. Symptomatic patients without evidence of viral pneumonia or hypoxia will be considered as mild cases.

Statistical analysis :

All data will be collected and analysed using Statistical Package for Social Science ( SPSS to investigate the incidence of liver injury at admission and its contribution to the development of AKI, severity of COVID-19 and outcomes in Sohag University hospital

Ethical Consideration :

The study will be assessed by scientific and ethical committee of Sohag faculty of medicine, an informed written consent will be obtained from all patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are positive for COVID-19 infection in Sohag University Hospital whose ages < 18 years old. (confirmed by polymerase chain reaction (PCR) from nasopharyngeal or oropharyngeal samples) who developed AKI at time of admission or during admission.

Exclusion Criteria:

* Patients whose ages >18 years old.
* Patients known to have any liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with respirator symptoms of COVID-19 admitted at Sohag university hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Relationship between liver enzymes and AKI in patients with COVID19 | 4 months
  Elevated Liver Enzymes as a predictor of Acute Kidney Injury in hospitalized patients with COVID-19

SECONDARY OUTCOMES:
Severity of COVID19 infection | 4 months
  Relationship between elevated liver enzymes and acute kidney injury as a predictor of Severity of COVID19

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ka Osman, Resident, Principal Investigator — Sohag university-faculty of medicine
Locations (1):
- SOHAGU, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol Methods Consent form
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April 2022 forever
Access Criteria: Any One have access

REFERENCES:
- [Background] Ngiam JN, Chew N, Tham SM, Lim ZY, Li TY, Cen S, Tambyah PA, Santosa A, Muthiah M, Sia CH, Cross GB. Elevated liver enzymes in hospitalized patients with COVID-19 in Singapore. Medicine (Baltimore). 2021 Jul 30;100(30):e26719. doi: 10.1097/MD.0000000000026719. PMID 34397705